CLINICAL TRIAL: NCT00172042
Title: A Study to Evaluate the Safety and Efficacy of Zoledronic Acid in the Prevention or Delaying of Bone Metastasis in Patients With Stage IIIA and IIIB Non-small Cell Lung Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Zoledronic Acid in the Prevention or Delaying of Bone Metastasis in Patients With Stage IIIA and IIIB Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CZOL446G2419
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2011-07-19 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; Bisphosphonates; Zoledronic acid; Bone metastases; Prevention of bone metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Zoledronic Acid

ARMS (2):
- Zoledronic acid (Experimental): Zoledronic acid 4 mg intravenous infusion over at least 15 minutes every 3 to 4 weeks for 24 months. Dosage was adjusted for participants with mild or moderate renal impairment.
  Interventions: Drug: Zoledronic acid 4 mg
- Control (Other): No investigational treatment. If a participant developed bone metastases, treatment was started with Zoledronic acid 4 mg intravenous infusion over at least 15 minutes every 3 to 4 weeks until 24 months from the date of study entry had elapsed.
  Interventions: Drug: Zoledronic acid 4 mg

INTERVENTIONS:
Drug: Zoledronic acid 4 mg — Zoledronic acid 4 mg in 5 mL concentrated solution prepared with 100 mL calcium free infusion solution (0.9 % sodium chloride or 5% glucose solution).
  Other Names: Zometa®

SUMMARY:
30-40% of patients with lung cancer will develop bone metastases during the course of their disease, which can lead to pain, decreased mobility and skeletal complications. This study will investigate the effect of zoledronic acid on preventing or delaying the development of bone metastases and the impact on disease progression/survival in patients with stage IIIA and IIIB Non-small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Non-small Cell Lung Cancer (NSCLC)
* Newly Diagnosed, Stage IIIA and Stage IIIB excluding patients with pleural effusion
* Patients must have received primary treatment for their disease and had no progression

Exclusion Criteria:

* Diagnosed with NSCLC longer than 6 months ago
* Treatment with other bisphosphonates in past 12 months
* Presence of metastases

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2005-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (69):
- Belgium (3):
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- China (3):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- France (2):
  - Novartis Investigative Site, Clamart
  - Novartis Investigative Site, Clémont
- Germany (14):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Ulm
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Patra - RIO
  - Novartis Investigative Site, Thessaloniki
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Mátraháza
  - Novartis Investigative Site, Pécs
- Italy (12):
  - Novartis Investigative Site, Bergamo
  - Novartis Investigative Site, Carpi
  - Novartis Investigative Site, Catania
  - Novartis Investigative Site, Como
  - Novartis Investigative Site, Cosenza
  - Novartis Investigative Site, Livorno
  - Novartis Investigative Site, Novara
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Reggio Calabria
  - Novartis Investigative Site, Rome
  - Novartis Investigative Site, Taormina
- Netherlands (4):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Hoofddorp
- Poland (4):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Seoul, South Korea
- Spain (5):
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Sabadell
- Taiwan (3):
  - Novartis Investigative Site, Lin-Ko
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chaingmai
- United Kingdom (6):
  - Novartis Investigative Site, Aberdeen
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Sutton

REFERENCES:
- [Derived] Scagliotti GV, Kosmidis P, de Marinis F, Schreurs AJM, Albert I, Engel-Riedel W, Schallier D, Barbera S, Kuo HP, Sallo V, Perez JR, Manegold C. Zoledronic acid in patients with stage IIIA/B NSCLC: results of a randomized, phase III study. Ann Oncol. 2012 Aug;23(8):2082-2087. doi: 10.1093/annonc/mds128. Epub 2012 Jun 22. PMID 22730101

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoledronic Acid | Control
Started | 226 | 211
Completed | 68 | 86
Not Completed | 158 | 125
Not completed — Adverse Event | 27 | 13
Not completed — Abnormal laboratory value(s) | 5 | 1
Not completed — Abnormal test procedure(s) | 0 | 3
Not completed — Unsatisfactory therapeutic effect | 13 | 11
Not completed — Patient no longer requires study drug | 10 | 8
Not completed — Protocol Violation | 8 | 7
Not completed — Withdrawal by Subject | 37 | 25
Not completed — Lost to Follow-up | 3 | 5
Not completed — Administrative problems | 13 | 10
Not completed — Death | 42 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Control | Total
Number analyzed (Participants) | 226 | 211 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.19) | 60.0 (9.27) | 59.6 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 65 | 130
  Male | 161 | 146 | 307

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-free survival is defined as the time from randomization to the date of the first documented progression or recurrence of disease or death from any cause. Time to disease progression (TTP) was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines with evaluations every 3 months.
Time Frame: Up to 24 months
Population: Intent-to-Treat Population consisting of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 226 | 211
Months | 9.0 [6.8 to 12.4] | 11.3 [7.7 to 15.8]

2. Secondary Outcome: Percentage of Participants With Bone Metastases at 6, 12, 18, and 24 Months
Description: Percentage of participants developing at least 1 bone metastasis, whether or not symptomatic. Bone scans were scheduled at screening and at 6-monthly intervals after study entry, or when symptoms suggested the presence of bone metastases. Positive bone scans required confirmation by x-ray, magnetic resonance imaging (MRI), or computed tomography (CT).
Time Frame: Months 6, 12, 18 and 24
Population: Intent-to-Treat Population consisting of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 226 | 211
Percentage of participants
  6 months | 2.2 [0.4 to 5.1] | 4.3 [0.0 to 4.0]
  12 months | 4.0 [1.1 to 7.3] | 7.1 [4.3 to 13.7]
  18 months | 6.2 [5.4 to 16.8] | 8.1 [6.9 to 18.3]
  24 months | 6.6 [6.2 to 18.5] | 9.0 [7.7 to 19.7]

3. Secondary Outcome: Kaplan-Meier Estimate of the Time to Occurrence of Bone Metastases
Description: Time to occurrence of bone metastases was defined as the time from randomization to the date of the first documented bone metastases which could be asymptomatic or symptomatic at the time of detection. Bone scans were scheduled at screening and at 6-monthly intervals after study entry, or when symptoms suggested the presence of bone metastases. Positive bone scans required confirmation by x-ray, magnetic resonance imaging (MRI), or computed tomography (CT).
Time Frame: Months 6, 12, 18, and 24
Population: Intent-to-Treat Population consisting of all randomized participants. Any participant without documented bone metastases at the date of analysis was to be censored at the date of the last bone scan.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 226 | 211
Percentage of participants
  6 months | 2.7 [0.4 to 5.1] | 1.9 [0.0 to 4.0]
  12 months | 4.2 [1.1 to 7.3] | 9.0 [4.3 to 13.7]
  18 months | 11.1 [5.4 to 16.8] | 12.6 [6.9 to 18.3]
  24 months | 12.4 [6.2 to 18.5] | 13.7 [7.7 to 19.7]

4. Secondary Outcome: Percentage of Participants With Skeletal Related Events (SREs) at 12 and 24 Months From Study Entry
Description: Skeletal Related Events were defined as radiation therapy or surgery to bone, spinal cord compression event or a pathologic bone fracture event.
Time Frame: Months 12 and 24
Population: Intent-to-Treat Population consisting of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 226 | 211
Percentage of participants
  12 months | 2.2 | 1.4
  24 months | 2.2 | 1.4

5. Secondary Outcome: Kaplan-Meier Estimates of the Time to the First Skeletal Related Event (SRE)
Description: Time to the first skeletal related event defined as the time from randomization to the date of occurrence of the first SRE. Skeletal Related Events were defined as radiation therapy or surgery to bone, spinal cord compression event or a pathologic bone fracture event
Time Frame: Months 6,12, 18, and 24
Population: Intent-to-Treat Population consisting of all randomized participants. Any participant in whom no SRE had been observed during the study was to be censored at the date of the last visit or the date of death whichever was the earlier.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 226 | 211
Percentage of participants
  6 month | 1.0 [0.0 to 2.3] | 0.0 [0.0 to 0.0]
  12 month | 2.7 [0.4 to 5.0] | 1.8 [0.0 to 3.9]
  18 month | 2.7 [0.4 to 5.0] | 1.8 [0.0 to 3.9]
  24 month | 2.7 [0.4 to 5.0] | 1.8 [0.0 to 3.9]

6. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival
Time Frame: Months 6, 12, 18, and 24
Population: Intent-to-Treat Population consisting of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 226 | 211
Percentage of participants
  6 months | 92.8 [88.4 to 95.5] | 93.6 [89.3 to 96.3]
  12 months | 81.8 [76.0 to 86.4] | 81.8 [75.7 to 86.5]
  18 months | 72.4 [65.7 to 78.0] | 71.0 [64.0 to 76.9]
  24 months | 59.5 [51.9 to 66.2] | 63.6 [56.1 to 70.1]

7. Primary Outcome: Kaplan-Meier Estimates for Progression-free Survival
Description: as for outcome 1
Time Frame: Months 6, 12, 18, and 24
Population: Intent-to-Treat Population consisting of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 226 | 211
Percentage of participants
  6 months | 63.0 [56.2 to 69.0] | 67.9 [61.0 to 73.9]
  12 months | 44.4 [37.6 to 51.0] | 48.8 [41.6 to 55.5]
  18 months | 30.7 [24.4 to 37.2] | 40.6 [33.7 to 47.5]
  24 months | 25.7 [19.8 to 32.0] | 36.0 [29.2 to 42.8]

8. Primary Outcome: Percentage of Participants With Progression-Free Survival Events
Description: Percentage of Participants with the Progression-free survival events: disease progression and death. Time to disease progression (TTP) was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines with evaluations every 3 months.
Time Frame: Up to 24 months
Population: Intent-to-Treat Population consisting of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Zoledronic Acid | Control
Number analyzed (Participants) | 226 | 211
Percentage of participants
  Disease Progression | 60.2 | 55.5
  Death | 8.4 | 5.7

ADVERSE EVENTS:
Description: Safety results are subsequently presented according to treatment actually received at the start of the study (224 in zoledronic acid arm, 213 in control arm); two patients were randomized to the zoledronic acid arm but did not receive study drug at the start of the study hence included into control arm for safety analysis.
Arm/Group | Zoledronic Acid | Control
Serious Adverse Events (participants affected / at risk) | 71/224 | 84/213
Other Adverse Events (participants affected / at risk) | 166/224 | 139/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=224) | Control (N=213)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiopulmonary failure (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 2 | 2
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastropleural fistula (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 4
Disease progression (General disorders) | 2 | 4
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 4 | 2
Influenza like illness (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 4
Sudden death (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Dental fistula (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 10
Post procedural infection (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 10
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 3 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Disorientation (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Labile blood pressure (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 2
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=224) | Control (N=213)
Anaemia (Blood and lymphatic system disorders) | 23 | 23
Abdominal pain upper (Gastrointestinal disorders) | 12 | 7
Constipation (Gastrointestinal disorders) | 32 | 13
Diarrhoea (Gastrointestinal disorders) | 12 | 13
Nausea (Gastrointestinal disorders) | 24 | 23
Vomiting (Gastrointestinal disorders) | 20 | 9
Asthenia (General disorders) | 11 | 15
Chest pain (General disorders) | 28 | 19
Fatigue (General disorders) | 38 | 26
Influenza like illness (General disorders) | 12 | 3
Pyrexia (General disorders) | 46 | 22
Bronchitis (Infections and infestations) | 6 | 11
Nasopharyngitis (Infections and infestations) | 17 | 19
Respiratory tract infection (Infections and infestations) | 15 | 12
Upper respiratory tract infection (Infections and infestations) | 7 | 16
Weight decreased (Investigations) | 11 | 12
Decreased appetite (Metabolism and nutrition disorders) | 31 | 29
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 11
Dizziness (Nervous system disorders) | 15 | 13
Headache (Nervous system disorders) | 19 | 23
Insomnia (Psychiatric disorders) | 21 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 60 | 54
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 49
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Rash (Skin and subcutaneous tissue disorders) | 17 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.